CLINICAL TRIAL: NCT03484130
Title: Prospective Phenotyping of Autonomous Aldosterone Secretion: A Cohort Study
Brief Title: Prospective Phenotyping of Autonomous Aldosterone Secretion
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Anand Vaidya, Director, Center for Adrenal Disorders, Brigham and Women's Hospital
Other Study IDs: 2018P000257
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Aldosterone Disorder; Adrenal Gland Disease; Blood Pressure
Keywords: primary aldosteronism
MeSH Terms: conditions — Adrenal Gland Diseases; Hyperaldosteronism | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High-Risk Normotensives: These high-risk normotensives are considered to be enriched for subclinical autonomous aldosterone secretion and have a high risk for developing incident hypertension
  Interventions: Dietary Supplement: Sodium loaded diet; Dietary Supplement: Restricted sodium diet

INTERVENTIONS:
Dietary Supplement: Sodium loaded diet — At baseline, and annually, participants will undergo aldosterone dynamic testing after ~5 days of a sodium loaded diet. The diet will consist of >180 mmol/day of sodium, ~50 mmol/day of potassium, and 600mg/d of calcium.
Dietary Supplement: Restricted sodium diet — At baseline, and annually, participants will undergo aldosterone dynamic testing after ~5 days of a sodium restricted diet. The diet will consist of <40 mmol/day of sodium, ~50 mmol/day of potassium, and 600mg/d of calcium.

SUMMARY:
This prospective cohort study will investigate the physiology and progression of autonomous aldosterone secretion.

DETAILED DESCRIPTION:
Primary aldosteronism is a disorder wherein aldosterone is secreted by the adrenal gland(s) independent of its physiologic regulators and cannot be appropriately suppressed with sodium/volume loading. Primary aldosteronism is a common cause of hypertension and has a relatively high prevalence. This is important since the excessive mineralocorticoid receptor activation in primary aldosteronism contributes to adverse cardiovascular and renal outcomes and death. For these reasons, it is critical that autonomous aldosteronism be detected early in its course since appropriate treatment interventions may prevent cardiovascular disease.

In addition to severe and overt primary aldosteronism in hypertension, human studies have shown that milder forms of primary aldosteronism can exist even among normotensive individuals. Detailed physiologic studies have shown that normotensive individuals with a phenotype of autonomous aldosterone secretion have greater cardiometabolic risk factors, impaired renal-vascular function, and a higher risk for developing incident hypertension. Further, older age is associated with greater autonomous aldosterone secretion, suggesting that autonomous aldosterone secretion may progress over time. A better understanding of the prevalence and progression of this type of "subclinical" autonomous aldosterone secretion may inform our understanding of the pathogenesis of hypertension and cardiometabolic diseases.

This protocol is designed to be a prospective longitudinal study that will carefully characterize the degree of autonomous aldosterone secretion among high-risk normotensive individuals and follow them longitudinally with repeated phenotyping study visits to assess the progression and severity of autonomous aldosterone secretion over time and its relevance to cardiovascular health. Phenotyping visits will include measurements of the renin-angiotensin-aldosterone system under controlled posture and variable sodium intakes and repeated assessments of blood pressure.

This prospective cohort study will provide insights into normal and abnormal aldosterone physiology over time and how it may contribute to time- or age-dependent hypertension and cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-70 years
2. Systolic blood pressure of 120-135 mmHg and/or diastolic blood pressure of 75-85 mmHg
3. At least one, or more, of the following:

   * BMI ≥ 25 kg/m2
   * Family history of hypertension prior to the age of 60 years in a parent or sibling
   * Diabetes with a hemoglobin A1c < 9%
4. If systolic blood pressure 115-135 mmHg and/or diastolic blood pressure 70-85 mmHg, must have two or more of the following:

   * BMI ≥ 25 kg/m2
   * Family history of hypertension prior to the age of 60 years in a parent or sibling
   * Diabetes with a hemoglobin A1c < 9%

Exclusion Criteria:

* Known history of hypertension or use of antihypertensive medications
* Known history of stroke, coronary artery disease, myocardial infarction, heart failure, cerebral or aortic aneurysm, or preeclampsia.
* Active cancer that is being treated with chemotherapeutic agents
* Pregnancy
* Breast feeding
* Daily use of prescribed opioid medications
* Illicit drug use (cocaine, heroin, methamphetamine)
* Daily non-steroidal anti-inflammatory medication use
* Daily use of glucocorticoids
* Electrocardiogram that shows evidence of prior myocardial infarction, atrial arrhythmia, left or right bundle branch blocks.
* Estimated glomerular filtration rate < 60 mL/min/1.73m2
* Active and untreated hyper- or hypo-thyroidism
* Abnormal screening laboratories (comprehensive metabolic panel, complete blood count, thyrotropin)
* BMI ≥ 45 kg/m2

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normotensive individuals who have a reasonably high risk of developing hypertension in the next few years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in renin | 10 years
  The primary outcome is to evaluate the longitudinal change in plasma renin activity

SECONDARY OUTCOMES:
SASSI | 5 years
  The longitudinal change in the sodium modulated suppression-to-stimulation index
Blood pressure | 5 years
  Longitudinal changes in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided